CLINICAL TRIAL: NCT04260776
Title: A SMART Pilot of Adaptive Treatment Strategies to Improve Engagement With a Web-Based Intervention for Socially Anxious Smokers
Brief Title: Adaptive Treatment Strategies for Improving Engagement With a Web-Based Smoking Intervention in Socially Anxious Smokers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI departure
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: RG1006869; NCI-2020-00302 (Registry Identifier: NCI / CTRP); K23DA048181 (NIH); 10384 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-06

CONDITIONS: Social Anxiety Disorder; Tobacco Use Disorder
MeSH Terms: conditions — Phobia, Social; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Participants will be randomly assigned to one of the two text message programs that correspond with the web-based intervention (MyWebQuit): 1) standard, 1-way text messages, or 2) interactive, 2-way text messages
  Interventions: Behavioral: Phase 1: Web-based intervention (MyWebQuit) with 1-way text messages; Behavioral: Phase 1: Web-based intervention (MyWebQuit) with interactive, 2-way text messages
- Phase 2 (Experimental): For the first 5 weeks after randomization, engagement with the website will be monitored. Participants who continue to engage with the website will continue with the same Phase 1 treatment components until the 3-month follow-up.
  Participants who disengage with the website will be randomly assigned to receive one of three re-engagement strategies: 1) interactive, re-engagement text messages, 2) re-engagement email, or 3) no re-engagement strategy
  Interventions: Behavioral: Phase 2: re-engagement text messages; Behavioral: Phase 2: re-engagement emails

INTERVENTIONS:
Behavioral: Phase 1: Web-based intervention (MyWebQuit) with 1-way text messages — Participants will receive MyWebQuit (web-based smoking intervention) along with a corresponding 1-way text messages
  Arms: Phase 1
Behavioral: Phase 1: Web-based intervention (MyWebQuit) with interactive, 2-way text messages — Participants will receive MyWebQuit (web-based smoking intervention) along with corresponding interactive, 2-way text messages
  Arms: Phase 1
Behavioral: Phase 2: re-engagement text messages — In addition to Phase 1 intervention components, 1/3 of participants who disengage with the website will receive interactive text messages designed to promote re-engagement
  Arms: Phase 2
Behavioral: Phase 2: re-engagement emails — In addition to Phase 1 intervention components, 1/3 of participants who disengage with the website will receive a personalized email designed to promote re-engagement
  Arms: Phase 2

SUMMARY:
This phase I trial will use a pilot sequential multiple assignment randomized trial (SMART) to examine protocol feasibility and acceptability of new components of a web-based intervention for socially anxious smokers. This study will be used to help build an adaptive treatment strategy to improve engagement with and effectiveness of the web-based intervention. Adaptive treatment strategies provide individualized sequences of intervention components to accommodate the changing needs of individuals based on their characteristics, treatment response, or engagement.

DETAILED DESCRIPTION:
This study proposes to use a pilot SMART to help build an adaptive treatment strategy to improve engagement with and effectiveness of a web-based intervention for socially anxious smokers. At the outset of the study (Phase 1), participants will receive access to a new web-based smoking intervention (MyWebQuit) and will randomized to receive one of two text message services: 1) 1-way text messages, or 2) interactive, 2-way text messages. Those who disengage with the website in the first 5 weeks will be re-randomized to one of three re-engagement strategies: 1) re-engagement emails, 2) re-engagement interactive text messages, or 3) no re-engagement strategy. Outcomes include protocol feasibility, treatment acceptability, treatment utilization, and smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* resides in the US and anticipates remaining in the US for the duration of the study
* smokes at least 5 cigarettes per day for at least 12 months prior to screening
* desire to quit smoking within 30 days
* has at least weekly internet access
* current use of a personal email account
* current use of text messaging
* willing to receive text messages as part of this study
* screen positive for social anxiety (LSAS-SR ≥ 60)
* interested in participating in the study for themselves (versus [vs] someone else)
* not currently taking part in any other smoking cessation treatment such as the nicotine patch, nicotine gum, Zyban, in-person counseling, telephone counseling, using a web-based or app-based cessation program
* no prior participation in one of the investigator's prior smoking cessation studies,
* comfortable reading, writing, and speaking English
* agree to the conditions of compensation
* not currently incarcerated in a prison
* willing to use the MyWebQuit program, complete study assessments, and sign an online consent form
* no other member of their same household participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Recruitment
  Number of individuals screened, eligible, consented; reasons for ineligibility
Data retention | 3 months
  Percentage of participants who complete outcome assessment at 3-months
Acceptability of intervention and Phase 1 engagement components | 3 months
  Treatment satisfaction ratings of the Phase 1 treatment conditions.
Acceptability of intervention and Phase 2 engagement components | 3 months
  Treatment satisfaction ratings of the Phase 2 treatment conditions
Utilization of interactive messages | 3 months
  Proportion of interactive text message prompts participants respond to
Utilization of Phase 1 text messages | 3 months
  Proportion of participants who unsubscribe from the Phase 1 text messages
Website Utilization | 3 months
  Total website logins
Website Utilization | 3 months
  Number of times disengagement criteria are met
Website Utilization | 3 months
  Percent of participants who login after rerandomization

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence abstinence | 3 months
  Preliminary efficacy for smoking cessation
Self-reported 30-day point prevalence abstinence | 3 months
  Preliminary efficacy for smoking cessation
Biochemically confirmed smoking abstinence | 3 months
  Preliminary efficacy for smoking cessation

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Watson, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No